CLINICAL TRIAL: NCT03908463
Title: KOMATE Registry: Korean Multicenter Angioplasty Team
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-0759
Record Dates: First submitted 2019-03-17; First posted 2019-04-09 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome; Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The patients who undergo percutaneous coronary intervention: The patients who undergo percutaneous coronary intervention will be enrolled.
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — All coronary intervention procedures will be performed according to current standard techniques.

SUMMARY:
The investigators will enroll the patients who underwent PCI and was based on real world clinical practice to collect the data regarding demographic, clinical, procedural information and clinical outcome using case report forms.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients older than 19 years
* 2. Patients who undergo percutaneous coronary intervention

Exclusion Criteria:

* 1. Refuse to participate
* 2. Pregnant women or women with potential childbearing

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients who undergo percutaneous coronary intervention group/Cohort Description: The patients who undergo percutaneous coronary intervention will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2018-10-05 (Actual); Primary Completion 2039-04 (Estimated); Study Completion 2039-04 (Estimated)

PRIMARY OUTCOMES:
Target lesion revascularization | Up to 20 years
  Defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLRs should be classified prospectively as clinically indicated or not clinically indicated by the investigator prior to repeat angiography. Clinically indicated revascularization: A revascularization is considered clinically indicated if angiography at followup shows a percent diameter stenosis ≥ 50% and if one of the following occurs:
  1. A positive history of recurrent angina pectoris, presumably related to the target vessel;
  2. Objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent), presumably related to the target vessel;
  3. Abnormal results of any invasive functional diagnostic test (eg, Doppler flow velocity reserve, fractional flow reserve);
  4. A TLR or TVR with a diameter stenosis ≥ 70% even in the absence of the above-mentioned ischemic signs or symptoms.
Target vessel revascularization | Up to 20 years
  Defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLRs should be classified prospectively as clinically indicated or not clinically indicated by the investigator prior to repeat angiography. Clinically indicated revascularization: A revascularization is considered clinically indicated if angiography at followup shows a percent diameter stenosis ≥ 50% and if one of the following occurs:
  1. A positive history of recurrent angina pectoris, presumably related to the target vessel;
  2. Objective signs of ischemia at rest (ECG changes) or during exercise test (or equivalent), presumably related to the target vessel;
  3. Abnormal results of any invasive functional diagnostic test (eg, Doppler flow velocity reserve, fractional flow reserve);
  4. A TLR or TVR with a diameter stenosis ≥ 70% even in the absence of the above-mentioned ischemic signs or symptoms.
Stent thrombosis | Up to 20 years
  Stent thrombosis is defined and discussed by the Academic Research Consortium
Myocardial infarction | Up to 20 years
  Myocardial Infarction Classification and Criteria for Diagnosis is defined by the Academic Research Consortium
Death | Up to 20 years
  All death will be recorded and their reason also be recorded. Also, cardiac death is defined as death due to myocardial infarction, cardiac perforation, tamponade, arrhythmia or any cardiac cause.
Non-target vessel revascularization | Up to 20 years
  Any revascularization of target-vessel revascularization will be collected.
Cerebrovascular accident | Up to 20 years
  Sudden onset of vertigo, numbness, aphasia, dysarthria or central neurologic deficit secondary to vascular lesions of the brain such as hemorrhage, embolism, thrombosis, or rupturing aneurysm, that persist for > 72 hours.
Major bleeding | Up to 20 years
  Any bleeding event will be collected with following description; the amount of hemoglobin drop or transfusion, the site of bleeding, any further treatment for the bleeding.
Cardiovascular readmission | Up to 20 years
  Any readmission due to cardiovascular adverse event will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Severance Cardiovascular Hospital Yonsei University College of Medicine, 250 Seongsanno, Seodaemun-gu 120-752 Seoul, South Korea, Seoul, South Korea

REFERENCES:
- [Derived] Cho S, Kang DY, Kim JS, Park DW, Kim IS, Kang TS, Ahn JM, Lee PH, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Lee SJ, Hong SJ, Ahn CM, Kim BK, Ko YG, Choi D, Jang Y, Hong MK, Park SJ. Dual antiplatelet therapy after percutaneous coronary intervention for left main coronary artery disease. Rev Esp Cardiol (Engl Ed). 2023 Apr;76(4):245-252. doi: 10.1016/j.rec.2022.07.007. Epub 2022 Jul 27. English, Spanish. PMID 35907438
- [Derived] Kim C, Kim JS, Kim H, Ahn SG, Cho S, Lee OH, Park JK, Shin S, Moon JY, Won H, Suh Y, Cho JR, Cho YH, Oh SJ, Lee BK, Hong SJ, Shin DH, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Jang Y. Consensus Decision-Making for the Management of Antiplatelet Therapy before Non-Cardiac Surgery in Patients Who Underwent Percutaneous Coronary Intervention With Second-Generation Drug-Eluting Stents: A Cohort Study. J Am Heart Assoc. 2021 Apr 20;10(8):e020079. doi: 10.1161/JAHA.120.020079. Epub 2021 Apr 10. PMID 33843258
- [Derived] Kim C, Kim JS, Kim H, Ahn SG, Cho S, Lee OH, Park JK, Shin S, Moon JY, Won H, Suh Y, Cho JR, Cho YH, Oh SJ, Lee BK, Hong SJ, Shin DH, Ahn CM, Kim BK, Ko YG, Choi D, Hong MK, Jang Y. Patterns of Antiplatelet Therapy During Noncardiac Surgery in Patients With Second-Generation Drug-Eluting Stents. J Am Heart Assoc. 2020 Jun 2;9(11):e016218. doi: 10.1161/JAHA.119.016218. Epub 2020 May 16. PMID 32419586